CLINICAL TRIAL: NCT00869206
Title: A Randomized, Phase III Study of Standard Dosing Versus Longer Dosing Interval of Zoledronic Acid in Metastatic Cancer
Brief Title: Zoledronic Acid in Treating Patients With Metastatic Breast Cancer, Metastatic Prostate Cancer, or Multiple Myeloma With Bone Involvement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CALGB-70604; CDR0000637947 (Registry Identifier: NCI Physician Data Query); NCI-2009-01102 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA037447 (NIH)
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Breast Adenocarcinoma; DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; Metastatic Malignant Neoplasm to the Bone; Pain; Musculoskeletal Complication; Urinary Complications
Keywords: pain; Prostate Adenocarcinoma; urinary complications; stage IV breast cancer; Recurrent Breast Carcinoma; stage IV prostate cancer; recurrent prostate cancer; Recurrent Prostate Carcinoma; stage I multiple myeloma; stage II multiple myeloma; Refractory Plasma Cell Myeloma; bone metastases
MeSH Terms: conditions — Pain; Breast Neoplasms; Prostatic Neoplasms; Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (zoledronic acid every 4 weeks) (Experimental): Patients receive zoledronic acid IV over at least 15 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: zoledronic acid
- Arm II (zoledronic acid every 12 weeks) (Experimental): Patients receive zoledronic acid IV over at least 15 minutes every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — Given IV

SUMMARY:
This randomized phase III trial studies two different schedules of zoledronic acid to compare how well they work in reducing bone-related complications in patients with breast cancer, prostate cancer, or multiple myeloma that has spread to other places in the body and have bone involvement. Bone-related complications are a major cause of morbidity in patients with metastatic prostate cancer, breast cancer, and multiple myeloma. Zoledronic acid may stop the growth of cancer cells in the bone and may help relieve some of the symptoms caused by bone metastases. It is not yet known whether giving zoledronic acid more or less frequently is more effective in treating patients with metastatic cancer that has spread to the bone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether every-12-week therapy with zoledronic acid is not inferior to every-4-week therapy for patients with metastatic breast cancer, metastatic prostate cancer, or multiple myeloma involving bone, as measured by the proportion who experience at least one skeletal related event within 24 months after randomization.

SECONDARY OBJECTIVES:

I. To compare pain scores (Brief Pain Inventory) of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing.

II. To compare the functional status (Eastern Cooperative Oncology Group [ECOG] performance status) of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing.

III. To compare the incidence of osteonecrosis of the jaw in patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing.

IV. To compare the incidence of renal dysfunction in patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing.

V. To compare the skeletal morbidity rate of these patients, defined as the number of skeletal-related events per year, of patients receiving every 12 week dosing to those receiving every 4 week dosing.

VI. To compare the suppression of serum markers of bone resorption of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing.

VII. To determine whether every 12 week therapy with zoledronic acid is not inferior to every-4-week therapy for each subgroup of patients with either breast cancer, prostate cancer, or multiple myeloma, as measured by the proportion who experience at least one skeletal related event within 24 months after randomization.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive zoledronic acid intravenously (IV) over at least 15 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive zoledronic acid IV over at least 15 minutes every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks for 2 years from registration.

ELIGIBILITY:
Eligibility Criteria:

* Histologic documentation of one of the following: breast adenocarcinoma, prostate adenocarcinoma or multiple myeloma
* At least one site of bone metastasis or bone involvement by radiologic imaging including plain radiograph, computed tomography (CT), positron emission tomography (PET) scan, PET/CT scan, magnetic resonance imaging, bone scan, or skeletal survey; indeterminate lesions should be confirmed by a second imaging method
* No prior treatment with IV bisphosphonates is allowed; prior treatment with oral bisphosphonates is allowed, but they must be discontinued prior to the initiation of protocol therapy
* No prior treatment with denosumab
* No prior treatment with radiopharmaceuticals; prior treatment with radioactive iodine is allowed; prostate cancer patients treated with brachytherapy are eligible
* Prior radiation therapy to bone is allowed, provided that at least one site of bone metastasis has not been irradiated and radiation is completed prior to registration; there should be no plan for radiation therapy to non-irradiated sites of bone metastases
* Prior adjuvant and metastatic chemotherapy, biologic therapy, and endocrine therapy is allowed
* No current treatment with investigational agent(s)
* Patients with known brain metastases are not eligible; patients who develop brain metastases during the study will be allowed to continue treatment as assigned
* Not pregnant and not nursing
* ECOG performance status 0-2
* Calculated creatinine clearance >= 30 mL/min
* Corrected serum calcium >= 8.0 mg/dL (2.00 mmol/L) and < 11.6 mg/dL (2.90 mmol/L) * Corrected serum calcium should be calculated using standard institutional practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1822 (Actual)
Dates: Start 2009-03; Primary Completion 2014-06 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L. Himelstein, MD, Study Chair — Helen F. Graham Cancer Center at Christiana Hospital
Locations (504):
- United States (503):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - North Bay Cancer Center, Fairfield, California
  - Valley Medical Oncology, Fremont, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Leavey Cancer Center at Northridge Hospital Medical Center, Northridge, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Feather River Hospital Cancer Center, Paradise, California
  - Pismo Beach, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Kaiser Permanente at Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Cancer Center of South Florida Foundation, Incorporated, Lake Worth, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Good Samaritan Hospital of Maryland, Baltimore, Maryland
  - Kaiser Permanente at Woodlawn Medical Center, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Kaiser Permanente - Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts Medical Center Cancer Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Quincy, Quincy, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Air Force Base Medical Center, Keesler Air Force Base, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates - Reno, Reno, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Trinitas Comprehensive Cancer Center at Trinitas Hospital, Elizabeth, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Medical Oncology and Hematology Associates of North Virginia - Fairfax, Fairfax, Virginia
  - Kaiser Permanente Medical Center - Fair Oaks, Fairfax, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Himelstein AL, Foster JC, Khatcheressian JL, Roberts JD, Seisler DK, Novotny PJ, Qin R, Go RS, Grubbs SS, O'Connor T, Velasco MR Jr, Weckstein D, O'Mara A, Loprinzi CL, Shapiro CL. Effect of Longer-Interval vs Standard Dosing of Zoledronic Acid on Skeletal Events in Patients With Bone Metastases: A Randomized Clinical Trial. JAMA. 2017 Jan 3;317(1):48-58. doi: 10.1001/jama.2016.19425. PMID 28030702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Started | 911 | 911
Completed | 882 | 884
Not Completed | 29 | 27

BASELINE CHARACTERISTICS:
Population: All baseline patients demographics were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks) | Total
Number analyzed (Participants) | 911 | 911 | 1822
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (12.1) | 65.3 (11.7) | 65.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 414 | 428 | 842
  Male | 497 | 483 | 980
Region of Enrollment [Number; unit: participants]
  United States | 911 | 911 | 1822

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Skeletal-related Event (SRE) Within 2 Years After Randomization
Description: To determine whether every-12-week therapy with zoledronic acid is not inferior to every-4-week therapy for patients with metastatic breast cancer, metastatic prostate cancer, or multiple myeloma involving bone, as measured by the proportion of patients who would have experienced at least one skeletal related event within 24 months after randomization.
Time Frame: 2 years
Population: All patients that were eligible and completed treatment were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Number analyzed (Participants) | 911 | 911
percentage of participants | 67.6 | 67.9
Statistical Analysis 1: Comparison: Arm I (Zoledronic Acid Every 4 Weeks) vs Arm II (Zoledronic Acid Every 12 Weeks); Test type: Non-Inferiority or Equivalence — Based on the published data on the effect of a standard of dosing schedule of > zoledronic acid compared to placebo, we choose ∆= 7%, πT= 42%, and πS= 35%. With a total of 1230 eligible patients (615 per arm), the probability of rejecting the null hypothesis using a one-sided test is at most 0.05 (Type I error α) when θ≥ 7% and the probability of rejecting the null hypothesis (the power) is at least 82% when θ≤0; p <= .05, Cochran-Mantel-Haenszel

2. Secondary Outcome: Average Pain Intensity Score as Assessed by the Brief Pain Inventory (BPI) Questionnaire
Description: To compare pain scores (Brief Pain Inventory) of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing. The change scores were evaluated in a general linear model with repeated measures for treatment effect and the time trend with patient-specific characteristics being adjusted for the mean interference score. Specifically the difference in score change per 4 weeks for Arm I using Arm II as the reference is reported. The score of the BPI questionnaire ranges from 0 being no pain to 10 being the most pain. The average score is reported for each arm below.
Time Frame: from baseline up to 2 years
Population: 1766 patients completed treatment and were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Number analyzed (Participants) | 882 | 884
score on a scale | 2.06 (0.14) | 2.09 (0.14)
Statistical Analysis 1: Comparison: Arm I (Zoledronic Acid Every 4 Weeks) vs Arm II (Zoledronic Acid Every 12 Weeks); Test type: Superiority or Other; p = 0.68, Mixed Models Analysis; Model is adjusted for tumor type, baseline creatinine, prior SREs, prior bisphosphonates, age, gender, race, BSA, and baseline performance status; Slope = -0.00394, Standard Error of Mean 0.009620

3. Secondary Outcome: Average ECOG Performance Status
Description: To compare functional status (ECOG performance status) of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing. The change scores were evaluated in a general linear model with repeated measures for treatment effect and the time trend with patient-specific characteristics being adjusted. Specifically the difference in score change per 4 weeks for Arm I using Arm II as the reference is reported. ECOG performance status is a measurement of a patients disability ranging from 0, fully active and able to carry out all pre disease performance without restriction, to 5, dead. The average performance status is reported below by arm.
Time Frame: from baseline up to 2 years
Population: 1766 patients completed treatment and were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Number analyzed (Participants) | 882 | 884
score on a scale | 0.82 (0.042) | 0.84 (0.042)
Statistical Analysis 1: Comparison: Arm I (Zoledronic Acid Every 4 Weeks) vs Arm II (Zoledronic Acid Every 12 Weeks); Test type: Superiority or Other; p = 0.64, Mixed Models Analysis; Adjusted for tumor type, baseline creatinine, prior SRE, prior bisphosphonates, age, gender, BSA, race, and baseline performance status; Slope = 0.0016, Standard Error of Mean 0.0034

4. Secondary Outcome: Incidence of Osteonecrosis of the Jaw
Description: To compare the incidence of osteonecrosis of the jaw in patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing. The percentage of participants with osteonecrosis is reported here.
Time Frame: from baseline up to 2 years
Population: 1766 patients completed treatment and were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Number analyzed (Participants) | 882 | 884
percentage of participants | 2.0 | 1.0

5. Secondary Outcome: Incidence of Renal Dysfunction
Description: To compare the incidence of renal dysfunction of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing. The percentage of patients with renal dysfunction, defined as grade 3 or grade 4 increased creatinine (Common Terminology Criteria for Adverse Events version 3.0), will be reported here.
Time Frame: from baseline up to 2 years
Population: 1689 patients completed treatment and were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Number analyzed (Participants) | 852 | 837
percentage of participants | 1.2 | .5
Statistical Analysis 1: Comparison: Arm I (Zoledronic Acid Every 4 Weeks) vs Arm II (Zoledronic Acid Every 12 Weeks); Test type: Superiority; p = 0.10, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.3 to 1.7]

6. Secondary Outcome: Skeletal Morbidity Rate
Description: To compare the skeletal morbidity rate, defined as the number of skeletal-related events per year, of patients receiving every 12 week dosing to those receiving every 4 week dosing.
Time Frame: from baseline up to 2 years
Population: 1766 patients were treated and analyzed.
Measure: Mean (Standard Deviation); unit: SRE's per year
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
Number analyzed (Participants) | 882 | 884
SRE's per year | .4 (1.0) | .4 (1.1)

7. Secondary Outcome: Bone Turnover Assessed by Serum C-telopeptide (CTX) Levels (Breast Cancer)
Description: To compare the suppression of serum markers of bone resorption of patients with metastatic breast cancer, metastatic prostate cancer, or myeloma involving bone receiving every 12 week dosing of zoledronic acid to those receiving every 4 week dosing. The number of patients with high & low CTX values by arm will be reported here.
Time Frame: from baseline up to 2 years
Population: 266 breast cancer patients who were treated and included in this portion of the substudy.
Measure: Count of Participants; unit: Participants
Groups:
- Breast Cancer 4 Weeks: Patients with Breast Cancer receive zoledronic acid IV over at least 15 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
- Breast Cancer 12 Weeks: Patients receive zoledronic acid IV over at least 15 minutes every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Breast Cancer 4 Weeks | Breast Cancer 12 Weeks
Number analyzed (Participants) | 137 | 129
Participants
  Low CTX (<0.415ng/ml) | 83 | 75
  High CTX (>0.415ng/ml) | 54 | 54

8. Secondary Outcome: Proportion of Patients Having at Least One SRE Within 24 Months After Randomization for the Subgroups of Patients With Breast Cancer
Description: To determine whether every 12 week therapy with zoledronic acid is not inferior to every-4-week therapy for patients with breast cancer, as measured by the proportion who experience at least one skeletal related event within 24 months after randomization.
Time Frame: from baseline up to 24 months
Population: 820 patients completed treatment and were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer 4 Weeks | Breast Cancer 12 Weeks
Number analyzed (Participants) | 410 | 410
Participants | 113 | 119

9. Secondary Outcome: Proportion of Patients Having at Least One SRE Within 24 Months After Randomization for the Subgroups of Patients With Prostate Cancer
Description: To determine whether every 12 week therapy with zoledronic acid is not inferior to every-4-week therapy for patients with prostate cancer, as measured by the proportion who experience at least one skeletal related event within 24 months after randomization.
Time Frame: from baseline up to 24 months
Population: 660 patients completed treatment and were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Prostate Cancer 4 Weeks: Patients with Prostate Cancer receive zoledronic acid IV over at least 15 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
- Prostate Cancer 12 Weeks: Patients with Prostate Cancer receive zoledronic acid IV over at least 15 minutes every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Prostate Cancer 4 Weeks | Prostate Cancer 12 Weeks
Number analyzed (Participants) | 330 | 330
Participants | 107 | 101

10. Secondary Outcome: Proportion of Patients Having at Least One SRE Within 24 Months After Randomization for the Subgroups of Patients With Multiple Myeloma
Description: To determine whether every 12 week therapy with zoledronic acid is not inferior to every-4-week therapy for patients with multiple myeloma, as measured by the proportion who experience at least one skeletal related event within 24 months after randomization.
Time Frame: from baseline up to 24 months
Population: 265 patient completed treatment and were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Multiple Myeloma 4 Weeks: Patients with Breast Cancer receive zoledronic acid IV over at least 15 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
- Multiple Myeloma 12 Weeks: Patients with Breast Cancer receive zoledronic acid IV over at least 15 minutes every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Multiple Myeloma 4 Weeks | Multiple Myeloma 12 Weeks
Number analyzed (Participants) | 130 | 135
Participants | 35 | 30

11. Secondary Outcome: Bone Turnover Assessed by Serum C-telopeptide (CTX) Levels (Prostate Cancer)
Description: as for outcome 7
Time Frame: from baseline up to 24 months
Population: 207 prostate cancer patients who were treated and included in this portion of the substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Cancer 4 Weeks | Prostate Cancer 12 Weeks
Number analyzed (Participants) | 104 | 103
Participants
  Low CTX (<0.415ng/ml) | 34 | 49
  High CTX (>.0.415ng/ml) | 70 | 54

12. Secondary Outcome: Bone Turnover Assessed by Serum C-telopeptide (CTX) Levels (Multiple Myeloma)
Description: as for outcome 7
Time Frame: from baseline up to 24 months
Population: 74 multiple myeloma patients were treated and included in this portion of the substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma 4 Weeks | Multiple Myeloma 12 Weeks
Number analyzed (Participants) | 38 | 36
Participants
  Low CTX (<0.415ng/ml) | 15 | 19
  High CTX (>.0.415ng/ml) | 23 | 17

ADVERSE EVENTS:
Arm/Group | Arm I (Zoledronic Acid Every 4 Weeks) | Arm II (Zoledronic Acid Every 12 Weeks)
All-Cause Mortality (participants affected / at risk) | 41/879 | 42/868
Serious Adverse Events (participants affected / at risk) | 96/879 | 103/868
Other Adverse Events (participants affected / at risk) | 779/879 | 750/868
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Zoledronic Acid Every 4 Weeks) (N=879) | Arm II (Zoledronic Acid Every 12 Weeks) (N=868)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (8) | 10 (11)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 3 (3) | 1 (2)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (2)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (2)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 12 (14)
Diarrhea (Gastrointestinal disorders) | 12 (13) | 11 (11)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (13) | 16 (17)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (9) | 9 (10)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 14 (14) | 14 (14)
Disease progression (General disorders) | 10 (10) | 15 (15)
Edema limbs (General disorders) | 1 (1) | 3 (4)
Fatigue (General disorders) | 6 (6) | 9 (10)
Fever (General disorders) | 3 (3) | 9 (9)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
General symptom (General disorders) | 1 (1) | 1 (2)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 3 (3) | 1 (1)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 4 (5)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative neurological injury - Spinal cord (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (3) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 9 (9) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin T increased (Investigations) | 2 (2) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 4 (4)
Lymphocyte count decreased (Investigations) | 4 (4) | 6 (6)
Neutrophil count decreased (Investigations) | 2 (2) | 6 (6)
Platelet count decreased (Investigations) | 5 (5) | 4 (4)
Weight loss (Investigations) | 2 (2) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 4 (6)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 28 (32) | 34 (39)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 7 (8) | 9 (10)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (5) | 11 (11)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (6) | 6 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 11 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 3 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 4 (5)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 23 (30) | 18 (22)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 9 (9)
Thrombosis (Vascular disorders) | 2 (4) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Zoledronic Acid Every 4 Weeks) (N=879) | Arm II (Zoledronic Acid Every 12 Weeks) (N=868)
Blood disorder (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (14) | 7 (8)
Hemoglobin decreased (Blood and lymphatic system disorders) | 98 (195) | 92 (206)
Hemolysis (Blood and lymphatic system disorders) | 16 (37) | 11 (29)
Lymphatic disorder (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 4 (5) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 3 (3) | 4 (4)
Cardiac pain (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 4 (4) | 3 (3)
Left ventricular failure (Cardiac disorders) | 7 (8) | 2 (3)
Myocardial ischemia (Cardiac disorders) | 7 (7) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 3 (8) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 1 (5)
Cushingoid (Endocrine disorders) | 1 (1) | 1 (2)
Endocrine disorder (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 4 (5) | 3 (3)
Diplopia (Eye disorders) | 1 (6) | 2 (3)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (2)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 4 (5) | 5 (23)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 2 (2)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 40 (74) | 42 (68)
Anal exam abnormal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 7 (15) | 1 (2)
Colitis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 348 (1527) | 333 (1341)
Dental prosthesis user (Gastrointestinal disorders) | 2 (5) | 2 (10)
Diarrhea (Gastrointestinal disorders) | 276 (693) | 275 (754)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 4 (25)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 6 (11)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 4 (4) | 2 (4)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (6) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4) | 4 (4)
Gingival pain (Gastrointestinal disorders) | 6 (9) | 6 (6)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 5 (6)
Nausea (Gastrointestinal disorders) | 367 (1187) | 357 (1069)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 7 (8) | 6 (15)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 5 (7)
Tooth development disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 6 (12)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 224 (441) | 198 (366)
Chest pain (General disorders) | 12 (14) | 19 (50)
Chills (General disorders) | 3 (4) | 0 (0)
Edema limbs (General disorders) | 16 (26) | 22 (51)
Facial pain (General disorders) | 4 (11) | 0 (0)
Fatigue (General disorders) | 90 (216) | 87 (260)
Fever (General disorders) | 173 (291) | 189 (298)
Flu-like symptoms (General disorders) | 2 (12) | 4 (4)
Gait abnormal (General disorders) | 4 (4) | 1 (1)
General symptom (General disorders) | 1 (1) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 97 (275) | 68 (157)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 4 (4)
Gallbladder obstruction (Hepatobiliary disorders) | 2 (3) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 4 (5) | 1 (6)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 3 (3) | 2 (2)
Bone infection (Infections and infestations) | 6 (6) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Catheter related infection (Infections and infestations) | 7 (11) | 2 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (2) | 1 (3)
Device related infection (Infections and infestations) | 0 (0) | 3 (3)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Ileal infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 12 (17) | 16 (20)
Joint infection (Infections and infestations) | 1 (2) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 16 (17) | 19 (20)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 13 (14) | 5 (5)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 5 (6) | 2 (3)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 19 (22) | 13 (14)
Uterine infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (3) | 1 (2)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 7 (8) | 14 (28)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Intraoperative musculoskeletal injury - Extremity-lower (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative neurological injury - NERVES: Sacral plexus (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
ADH abnormal (Investigations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 20 (27) | 14 (23)
Alkaline phosphatase increased (Investigations) | 46 (99) | 34 (80)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 39 (58) | 23 (29)
Blood bilirubin increased (Investigations) | 15 (17) | 12 (18)
Cardiac troponin I increased (Investigations) | 0 (0) | 2 (2)
Cardiac troponin T increased (Investigations) | 2 (2) | 0 (0)
Coagulopathy (Investigations) | 0 (0) | 2 (2)
Creatine phosphokinase increased (Investigations) | 2 (4) | 2 (2)
Creatinine increased (Investigations) | 14 (23) | 10 (10)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0)
INR increased (Investigations) | 8 (28) | 4 (18)
Laboratory test abnormal (Investigations) | 4 (6) | 0 (0)
Leukocyte count decreased (Investigations) | 68 (128) | 70 (160)
Lipase increased (Investigations) | 1 (1) | 2 (3)
Lymphocyte count decreased (Investigations) | 41 (126) | 45 (143)
Neutrophil count decreased (Investigations) | 79 (131) | 70 (118)
Platelet count decreased (Investigations) | 53 (108) | 59 (138)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 4 (24) | 6 (32)
Weight loss (Investigations) | 11 (27) | 14 (30)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 28 (48) | 24 (39)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 43 (150) | 57 (181)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 20 (23) | 22 (22)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (29)
Serum albumin decreased (Metabolism and nutrition disorders) | 22 (30) | 12 (18)
Serum calcium decreased (Metabolism and nutrition disorders) | 320 (996) | 290 (839)
Serum calcium increased (Metabolism and nutrition disorders) | 87 (177) | 82 (207)
Serum glucose decreased (Metabolism and nutrition disorders) | 4 (5) | 5 (9)
Serum magnesium increased (Metabolism and nutrition disorders) | 56 (101) | 61 (93)
Serum phosphate decreased (Metabolism and nutrition disorders) | 64 (95) | 69 (130)
Serum potassium decreased (Metabolism and nutrition disorders) | 30 (41) | 26 (45)
Serum potassium increased (Metabolism and nutrition disorders) | 11 (13) | 11 (12)
Serum sodium decreased (Metabolism and nutrition disorders) | 31 (45) | 28 (38)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 93 (307) | 83 (311)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (20) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 191 (792) | 177 (688)
Bone pain (Musculoskeletal and connective tissue disorders) | 139 (595) | 131 (452)
Buttock pain (Musculoskeletal and connective tissue disorders) | 24 (52) | 17 (32)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 25 (74) | 21 (39)
Fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 22 (27) | 19 (22)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (16) | 5 (8)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 (7) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 46 (73) | 44 (79)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 29 (58) | 38 (79)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 15 (20) | 5 (10)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 114 (318) | 92 (311)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 6 (6)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (4)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Arachnoiditis (Nervous system disorders) | 1 (3) | 0 (0)
Ataxia (Nervous system disorders) | 3 (3) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 15 (30) | 16 (27)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 2 (2) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 3 (9) | 0 (0)
Headache (Nervous system disorders) | 29 (58) | 37 (63)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 6 (6)
Memory impairment (Nervous system disorders) | 2 (4) | 1 (1)
Neuralgia (Nervous system disorders) | 4 (8) | 7 (8)
Neurological disorder NOS (Nervous system disorders) | 7 (10) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 17 (33) | 11 (18)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (91) | 51 (215)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis brachial (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 6 (7)
Sinus pain (Nervous system disorders) | 1 (2) | 2 (2)
Speech disorder (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 14 (20) | 11 (15)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (10) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (6) | 4 (5)
Confusion (Psychiatric disorders) | 4 (14) | 6 (6)
Depression (Psychiatric disorders) | 4 (6) | 12 (25)
Insomnia (Psychiatric disorders) | 6 (16) | 6 (11)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 2 (2) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 2 (2) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (3) | 0 (0)
Kidney pain (Renal and urinary disorders) | 3 (3) | 4 (4)
Kidney perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 2 (2)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 8 (13)
Urinary incontinence (Renal and urinary disorders) | 4 (19) | 2 (4)
Urinary retention (Renal and urinary disorders) | 4 (6) | 4 (4)
Urogenital disorder (Renal and urinary disorders) | 183 (794) | 159 (677)
Breast pain (Reproductive system and breast disorders) | 7 (42) | 10 (16)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 14 (31) | 9 (12)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Prostatic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (4)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (33)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 42 (71) | 51 (78)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 14 (14)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 13 (30)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (11) | 4 (8)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 12 (21) | 8 (39)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (13) | 7 (19)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 4 (6)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (13)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2) | 9 (32)
Hypertension (Vascular disorders) | 32 (75) | 21 (55)
Hypotension (Vascular disorders) | 8 (9) | 12 (12)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 23 (34) | 24 (47)
Vascular disorder (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days